CLINICAL TRIAL: NCT06035029
Title: Research on Intestinal Flora and Metabonomics of Appendicitis in Children
Brief Title: Intestinal Flora and Metabonomics of Appendicitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HongyiQu (Other)
Responsible Party: Sponsor-Investigator, HongyiQu, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023 （009）
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Appendicitis; Intestinal Metaplasia; Metabonomics
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Before antibiotics for children in the case group, a stool sample (5-10 g) was collected from all of the included subjects and placed in a sterile enzyme-free (no RNA and DNA enzyme) cryopreservation tube.
  When children with appendicitis are taken to the operating room and placed under anesthesia, the patient is collected and collected after storage using sterile preservation fluid. After the appendectomy, the full length of the appendix cavity was wiped with a sterile cotton swab under a sterile environment, and then the swab was placed into a sterile collection tube. Specimens were transported and stored at-80℃ until analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Children with appendectomy for appendicitis
- Control group: Children with no digestive disease or medical history

SUMMARY:
The goal of this observational study is to learn about the key bacterial flora and metabolites associated with appendicitis in children. The main questions it aims to answer are:

* To screen out the key biomarkers of pediatric appendicitis.
* What are the microbial differences in different parts of pediatric appendicitis patients.

Participants will detect feces using 16s ribosomal RiboNucleicAcid (16S rRNA) gene sequencing technology and differences of the fecal metabolites between healthy children and appendicitis children were analyzed using untargeted metabolomics based on Liquid chromatography-tandem mass spectrometry(LC-M S/MS) platform.Through the analysis of intestinal bacterial flora and metabolomics association and the differential analysis of intestinal bacterial flora in different parts of the case group, the key bacterial flora and metabolites were excavated.

DETAILED DESCRIPTION:
Participants will detect feces using 16s ribosomal RiboNucleicAcid (16S rRNA) gene sequencing technology and differences of the fecal metabolites between healthy children and appendicitis children were analyzed using untargeted metabolomics based on Liquid chromatography-tandem mass spectrometry(LC-M S/MS) platform.

Differences in the intestinal flora of different parts of the case group: the intestinal flora of the case group in feces and rectum were detected by 16s ribosomal RiboNucleicAcid (16S rRNA) gene sequencing technology, and the intestinal flora of different parts were analyzed and compared.

Through the analysis of intestinal bacterial flora and metabolomics association and the differential analysis of intestinal bacterial flora in different parts of the case group, the key bacterial flora and metabolites were excavated.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-14 years who were initially diagnosed with appendicitis and underwent laparoscopic appendectomy
* Children aged 1-14 years with non-digestive tract disease and no history of digestive tract disease

Exclusion Criteria:

* A family history of intestinal disease
* Allergic to antibiotic therapy drugs
* Patients with long-term drug use causing microbial structure changes or intestinal flora disorders
* Patients with other congenital diseases such as Meckel's diverticulum, intestinal rotation and other malrotation
* With other systemic diseases, such as obvious upper respiratory tract infection or myocarditis
* Children with other digestive system diseases after auxiliary examination or surgical diagnosis

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 1-14 in Department of Pediatric Surgery in Shandong Qianfoshan Hospital
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The 16S rRNA gene sequence | up to 24 weeks
  Samples were qualified for Polymerase Chain Reaction(PCR) amplification of the V3 and V4 variable regions of the 16 rRNA gene. The Polymerase Chain Reaction(PCR) products were then quantified by confirming the presence of PCR amplicons by gel electrophoresis on a 2% agarose gel and staining with ethidium bromide, and equimolar amounts (100 ng) of PCR amplicons were pooled prior to pyrosequencing. High-throughput sequencing of the qualified 16S amplicon libraries.
Fecal untargeted metabolomics testing | up to 24 weeks
  To analyze the fecal metabolite differences and the correlation of appendicitis and metabolites using untargeted metabolomics based on the LC-M S/MS platform. To screen key metabolites in pediatric appendicitis.

CONTACTS AND LOCATIONS:
Overall Officials: Qu, Study Chair — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital Of Shandong First Medcial Unversity, Jinan, Shandong, China